CLINICAL TRIAL: NCT00003835
Title: Phase III Intergroup Trial of Irinotecan (CPT-11) (NSC# 616348) Plus Fluorouracil/Leucovorin (5-FU/LV) Versus Fluorouracil/Leucovorin Alone After Curative Resection for Patients With Stage III Colon Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Stage III Colon Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: SWOG Cancer Research Network (Network); North Central Cancer Treatment Group (Network); Eastern Cooperative Oncology Group (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01844; NCI-2012-01844 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-C89803; NCCTG-C89803; CDR0000066992; CAN-NCIC-CO15; E-89803; CALGB 89803 (Other: Cancer and Leukemia Group B); C89803 (Other: CTEP); U10CA031946 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Adenocarcinoma of the Colon; Stage III Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Leucovorin; Fluorouracil; Irinotecan

ARMS (2):
- Arm I (leucovorin calcium and fluorouracil) (Experimental): Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV beginning 1 hour into leucovorin calcium infusion weekly for 6 weeks. Treatment is repeated every 8 weeks for 4 courses.
  Interventions: Drug: leucovorin calcium; Drug: fluorouracil; Other: laboratory biomarker analysis
- Arm II (leucovorin calcium, fluorouracil, irinotrcan) (Experimental): Patients receive irinotecan IV over 90 minutes, followed by leucovorin calcium IV, then followed by fluorouracil IV weekly for 4 weeks. Treatment is repeated every 6 weeks for 5 courses
  Interventions: Drug: leucovorin calcium; Drug: fluorouracil; Drug: irinotecan hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: leucovorin calcium — Given IV
Drug: fluorouracil — Given IV
Drug: irinotecan hydrochloride — Given IV
  Arms: Arm II (leucovorin calcium, fluorouracil, irinotrcan)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which chemotherapy regimen is more effective for stage III colon cancer. Randomized phase III trial to compare the effectiveness of fluorouracil plus leucovorin with or without irinotecan in treating patients who have undergone surgery for stage III colon cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the overall and disease free survival of patients with stage III colon cancer treated with adjuvant fluorouracil and leucovorin calcium with or without irinotecan.

II. Assess prognostic markers and correlate their expression with disease free and overall survival of these patients.

III. Assess the influence of diet, body mass index, and physical activity on the risk of cancer recurrence and survival in these patients.

IV. Assess the influence of diet, obesity, and physical activity on the risk of toxicity associated with adjuvant therapy in these patients.

V. Determine whether pathological features (including tumor grade, tumor mitotic (proliferation) index, tumor border configuration, and host lymphoid response to tumor; and lymphatic vessel, venous vessel and perineural invasion) predict outcome in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to lymph node involvement (1-3 vs 4 or more), histology (poorly differentiated or undifferentiated vs well or moderately differentiated), and preoperative serum CEA (less than 5.0 ng/mL vs at least 5.0 ng/mL vs unknown). Study therapy must begin within 21-56 days after surgery. Patients are randomized to one of two treatment arms:

ARM I: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV beginning 1 hour into leucovorin calcium infusion weekly for 6 weeks. Treatment is repeated every 8 weeks for 4 courses.

ARM II: Patients receive irinotecan IV over 90 minutes, followed by leucovorin calcium IV, then followed by fluorouracil IV weekly for 4 weeks. Treatment is repeated every 6 weeks for 5 courses.

Patients complete a food questionnaire at the beginning of the third course and then at 6 months after study therapy.

Patients are followed every 3 months for 2 years, every 4 months for 2 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 1260 patients will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented adenocarcinoma of the colon; the gross inferior (caudad) margin of the primary tumor must lie above the peritoneal reflection; tumor must have been completely resected, including negative radial resecting margins
* There must be no history of distant metastatic disease at the time of registration
* Pathological evaluation must show Modified Astler-Coller stage C (TxN1-2M0) disease
* No previous or concurrent malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for five years
* Zubrod performance status of 0-2
* Non-pregnant and not nursing, as chemotherapy is thought to present substantial risk to the fetus/infant; men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while in this study
* Granulocytes >= 1,500/ul
* Platelet count >= 100,000/ul
* Creatinine =< 1.5 x upper limits of normal
* Bilirubin =< upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1260 (Estimated)
Dates: Start 1999-05; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time to recurrence | From time of resection until documented disease progression, assessed up to 6 years
  The Cox proportional hazards model will be used to determine the association between each marker and time to recurrence and survival controlling for other baseline factors such as age, gender, treatment, primary tumor site, degree of differentiation.
Survival | Up to 6 years
  The Cox proportional hazards model will be used to determine the association between each marker and time to recurrence and survival controlling for other baseline factors such as age, gender, treatment, primary tumor site, degree of differentiation.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saltz, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States

REFERENCES:
- [Derived] Lee S, Ma C, Zhang S, Ou FS, Bainter TM, Niedzwiecki D, Saltz LB, Mayer RJ, Whittom R, Hantel A, Benson A, Atienza D, Kindler H, Gross CP, Irwin ML, Meyerhardt JA, Fuchs CS. Marital Status, Living Arrangement, and Cancer Recurrence and Survival in Patients with Stage III Colon Cancer: Findings from CALGB 89803 (Alliance). Oncologist. 2022 Jun 8;27(6):e494-e505. doi: 10.1093/oncolo/oyab070. PMID 35641198
- [Derived] Symonds L, Yu M, Zhang Y, Ou FS, Zemla TJ, Carter K, Bertagnolli M, Innocenti F, Bosch LJ, Meijer GA, Carvalho B, Grady WM, Cohen SA. Evaluation of methylated DCR1 as a biomarker for response to adjuvant irinotecan-based therapy in stage III colon cancer: cancer and leukaemia Group B 89803 (Alliance). Epigenetics. 2022 Dec;17(12):1715-1725. doi: 10.1080/15592294.2022.2058225. Epub 2022 Apr 12. PMID 35412430
- [Derived] Kosumi K, Hamada T, Zhang S, Liu L, da Silva A, Koh H, Twombly TS, Mima K, Morikawa T, Song M, Nowak JA, Nishihara R, Saltz LB, Niedzwiecki D, Ou FS, Zemla T, Mayer RJ, Baba H, Ng K, Giannakis M, Zhang X, Wu K, Giovannucci EL, Chan AT, Fuchs CS, Meyerhardt JA, Ogino S. Prognostic association of PTGS2 (COX-2) over-expression according to BRAF mutation status in colorectal cancer: Results from two prospective cohorts and CALGB 89803 (Alliance) trial. Eur J Cancer. 2019 Apr;111:82-93. doi: 10.1016/j.ejca.2019.01.022. Epub 2019 Mar 1. PMID 30826660
- [Derived] Van Blarigan EL, Ou FS, Niedzwiecki D, Zhang S, Fuchs CS, Saltz L, Mayer RJ, Venook A, Ogino S, Song M, Benson A, Hantel A, Atkins JN, Giovannucci EL, Meyerhardt JA. Dietary Fat Intake after Colon Cancer Diagnosis in Relation to Cancer Recurrence and Survival: CALGB 89803 (Alliance). Cancer Epidemiol Biomarkers Prev. 2018 Oct;27(10):1227-1230. doi: 10.1158/1055-9965.EPI-18-0487. Epub 2018 Jul 23. PMID 30038051
- [Derived] Van Blarigan EL, Fuchs CS, Niedzwiecki D, Zhang S, Saltz LB, Mayer RJ, Mowat RB, Whittom R, Hantel A, Benson A, Atienza D, Messino M, Kindler H, Venook A, Ogino S, Giovannucci EL, Ng K, Meyerhardt JA. Association of Survival With Adherence to the American Cancer Society Nutrition and Physical Activity Guidelines for Cancer Survivors After Colon Cancer Diagnosis: The CALGB 89803/Alliance Trial. JAMA Oncol. 2018 Jun 1;4(6):783-790. doi: 10.1001/jamaoncol.2018.0126. PMID 29710284
- [Derived] Fadelu T, Zhang S, Niedzwiecki D, Ye X, Saltz LB, Mayer RJ, Mowat RB, Whittom R, Hantel A, Benson AB, Atienza DM, Messino M, Kindler HL, Venook A, Ogino S, Ng K, Wu K, Willett W, Giovannucci E, Meyerhardt J, Bao Y, Fuchs CS. Nut Consumption and Survival in Patients With Stage III Colon Cancer: Results From CALGB 89803 (Alliance). J Clin Oncol. 2018 Apr 10;36(11):1112-1120. doi: 10.1200/JCO.2017.75.5413. Epub 2018 Feb 28. PMID 29489429
- [Derived] Fuchs MA, Yuan C, Sato K, Niedzwiecki D, Ye X, Saltz LB, Mayer RJ, Mowat RB, Whittom R, Hantel A, Benson A, Atienza D, Messino M, Kindler H, Venook A, Innocenti F, Warren RS, Bertagnolli MM, Ogino S, Giovannucci EL, Horvath E, Meyerhardt JA, Ng K. Predicted vitamin D status and colon cancer recurrence and mortality in CALGB 89803 (Alliance). Ann Oncol. 2017 Jun 1;28(6):1359-1367. doi: 10.1093/annonc/mdx109. PMID 28327908
- [Derived] Pavelitz T, Renfro L, Foster NR, Caracol A, Welsch P, Lao VV, Grady WB, Niedzwiecki D, Saltz LB, Bertagnolli MM, Goldberg RM, Rabinovitch PS, Emond M, Monnat RJ Jr, Maizels N. MRE11-deficiency associated with improved long-term disease free survival and overall survival in a subset of stage III colon cancer patients in randomized CALGB 89803 trial. PLoS One. 2014 Oct 13;9(10):e108483. doi: 10.1371/journal.pone.0108483. eCollection 2014. PMID 25310185
- [Derived] Ogino S, Liao X, Imamura Y, Yamauchi M, McCleary NJ, Ng K, Niedzwiecki D, Saltz LB, Mayer RJ, Whittom R, Hantel A, Benson AB 3rd, Mowat RB, Spiegelman D, Goldberg RM, Bertagnolli MM, Meyerhardt JA, Fuchs CS; Alliance for Clinical Trials in Oncology. Predictive and prognostic analysis of PIK3CA mutation in stage III colon cancer intergroup trial. J Natl Cancer Inst. 2013 Dec 4;105(23):1789-98. doi: 10.1093/jnci/djt298. Epub 2013 Nov 14. PMID 24231454
- [Derived] Yothers G, Sargent DJ, Wolmark N, Goldberg RM, O'Connell MJ, Benedetti JK, Saltz LB, Dignam JJ, Blackstock AW; ACCENT Collaborative Group. Outcomes among black patients with stage II and III colon cancer receiving chemotherapy: an analysis of ACCENT adjuvant trials. J Natl Cancer Inst. 2011 Oct 19;103(20):1498-506. doi: 10.1093/jnci/djr310. Epub 2011 Oct 12. PMID 21997132
- [Derived] McCleary NJ, Niedzwiecki D, Hollis D, Saltz LB, Schaefer P, Whittom R, Hantel A, Benson A, Goldberg R, Meyerhardt JA. Impact of smoking on patients with stage III colon cancer: results from Cancer and Leukemia Group B 89803. Cancer. 2010 Feb 15;116(4):957-66. doi: 10.1002/cncr.24866. PMID 20052723